CLINICAL TRIAL: NCT05485623
Title: The Use of PulseNmore FC Device in Patients Undergoing IVF Treatment A Study to Evaluate the Safety and the Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: PulseNmore (Industry)
Responsible Party: Principal Investigator, YoelShufaro, Head of IVF Unit, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0271-21
Record Dates: First submitted 2022-07-14; First posted 2022-08-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Women Undergoing Fertility Treatments

STUDY DESIGN:
Intervention Model Description: Approximately 120 women will be recruited to accommodate 20% drop out. A comparison between FC scan and in-clinic scan (ground truth - GT) will be performed in order to assess the safety, feasibility and efficacy of the Pulsenmore FC device in the two operation modes.
  Naïve subjects who haven't use the FC device will be allocated to use the CG-mode. While experienced patients who already used the FC device will be offered to use the AG mode for a second cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinician guided scan comparing the device output to the in clinic scan (ground truth) (Experimental): Naïve subjects who haven't use the FC device will be allocated to use the CG-mode
  The patient will perform a CG scan, guided by a professional sonographer on a Pulsenmore telehealth platform, who will instruct the patient during the exam. At visit 1: the procedure will be performed in a private room in the clinic, while the clinician will be in a different room than the patient. At visit 2 and all other visits, until the last visit, FC scans will be done from home. The clinician will guide the patient using a standardized language which was practiced and used during the clinician training. By the end of the scan, the patient will transmit the videos to the cloud. Then the clinician will review the video scans for visualization of ovaries and uterus, identifying the number and size of ovarian follicles, endometrial thickness and additional parameters
  Interventions: Device: PulseNmore FC
- App guided scan comparing the device output to the in clinic scan (ground truth) (Experimental): Experienced patients who already used the FC device will be offered to use the AG node for a second cycle.
  The patient will perform self - administered vaginal sonography using the study device and assisted by videos on Pulsenmore app. The procedure will be performed at home, in the morning before the patient come to the clinic for the conventional US and tests. All scans are automatically uploaded to the Pulsenmore web-viewer. A qualified reviewer will review the videos for visualization of ovaries and uterus, identify the number and size of ovarian follicles, and measure endometrial thickness. Other parameters might be evaluated as well. The App guided scan is limited to 4 minutes and the session will be deactivated by the end of the scanning time.
  Interventions: Device: PulseNmore FC

INTERVENTIONS:
Device: PulseNmore FC — Pulsenmore Ltd. has developed a small portable vaginal ultrasound device for personal use at home. The ultrasound device allows to scan and assess both the uterus and the ovaries. This ultrasound device connects to a smartphone and a user-friendly application simplifies its use. This ultrasound device is based on the company's 'Pulsenmore ES ultrasound system' which is a small abdominal ultrasound device for home and self-use by pregnant women. This (abdominal) ultrasound device allows scanning and detection of fetal pulse, count fetal movements, assess the amount of amniotic fluid and more. The device is an abdominal ultrasound probe that connects to a smartphone using a specially designed socket. The main difference between the devices is the different design of the ultrasound vaginal probe.
  The device consists of 2 components: a cradle and an application (software). The cradle contains the electronic components and the ultrasound probe.

SUMMARY:
This is a single center, interventional, longitudinal prospective, of 100 women undergoing fertility treatment in the IVF unit of Belinson Hospital. The study will examine the performance of the FC Clinician-Guided (CG) transvaginal scan done with Pulsenmore FC device, performed by patients with remote guidance of a professional sonographer. Experienced patients who already used the FC device for one cycle in a CG mode, can be re-enrolled for testing also the App-Guided mode of the device. All FC scans will be compared to the conventional ultrasound system in-clinic scan (ground truth - GT). Subjects will participate in the study for one IVF cycle (or 2 cycles if patient is re-enrolled also for the APP mode), an estimated study period of 2 weeks, and scan schedule protocol will follow the standard of care scan schedule for IVF treatment. The last visit will be defined when the attending physician concludes that the follicle requitement potential of the cycle has been achieved and the patient is ready for oocyte aspiration.

DETAILED DESCRIPTION:
1. The primary safety endpoint for each study subject is whether there is severe device- or procedure- related adverse events observed during the study. The resulting event rates will be established separately for the video guided and clinician guided modes of the device.
2. Primary Effectiveness Endpoints. The study will examine the performance of the clinician guided modes of the device. This shall be utilizing various parameters in acquired images/clips utilizing the Pulsenmore FC system, "the candidate device", in the:

Clinician guided mode- the self-transvaginal scan is performed by the patient with the remote guidance of a professional sonographer.

Comparing them to the conventional ultrasound system in clinical settings (ground truth - GT) in terms of visualization of the ovaries and uterus. The study will be considered successful for video guided and clinician guided separately, based on the concordance level of visualization of the ovaries and uterus when compared to GT in each visit and at the last visit.

Study target population: 100 women ages 18-43 undergoing ovarian stimulation in the IVF unit of Belinson Hospital.

For CG mode evaluation - naive subjects, who have never used the FC device. For AG mode evaluation - Subjects who participate in the study and have already used the FC device in a CG mode for one cycle.

Study Design Summary: This is a single centre, longitudinal investigational prospective study, of 100 women undergoing fertility treatment in the IVF unit of Belinson Hospital. A comparison between FC scan and in-clinic scan (ground truth - GT) will be performed in order to assess the safety, feasibility and efficacy of the Pulsenmore FC device in the two operation modes.

Study subjects will each perform a total of 5-6 ultrasound visits. The number of visits will be determined by the treating physician according to the IVF cycle progression.

Subject will undergo screening and Inform consent process. Then, patient will receive FC device and phone to be used during the study. The training and qualification will be done via the CG mode, with the goal to confirm the patient's physical suitability, capability and willing to participate the study.

Following training, patient will undergo her first US sessions: first the CG scan and then the in-clinic scan. Only at visit 1 both scanning sessions will be performed at the clinic by the clinic' sonographer. Then, the patient will take the FC device & phone to be used at home at the next visits.

Each visit constituting of 2 different scans (CG or AG and in-clinic scan). During the ART cycle, the scan schedule protocol will follow the standard of care scan schedule for ovary stimulation treatment.

FC scans will be done remotely, at the patient's home in the morning. The FC sessions will be done at the same day and before the in-clinic visit. CG scan will be guided by an external sonographer. AG scan will be done by the patient with no guidance. The in-clinic US session will be performed in the clinic at the same morning, by the clinic's sonographer, no later than 3 hours after the CG session.

The last study visit is the visit before trigger and before Ovary Pick-UP (OPU). The patient will return the device and phone when she comes to the clinic for the OPU procedure.

Following completion of the last visit, patient and sonographer will receive an online questionnaire for evaluation their satisfaction and user experience as well as the subject capability to use AG mode in the next cycle, if relevant.

Before the enrolment of the 100 patients begins, a pilot study of 4 patients, 2 in each application mode which will follow the same protocol will be enrolled. The purpose of the pilot is to streamline the procedure. They will be included in the safety outcome of the study but will not be part of the effectiveness determination of the product. The enrolment of the 100 patients will begin after the 4 initial patients were completed.

Scans reading and interpretation:

All results from the App guided scan/ clinician guided scan and in-clinic scans will be stored and compared. If any discordant data is found, additional independent reviewer, acquired by the company will read the scans in question. The in-clinic scan will be used as the gold standard. The independent reviewers should be blinded to the in-clinic scan and to the previous device output scans. Majority rule (two of three) will be used to establish the correct reading of any of the discordant parameters in the video guided and clinician guided modes.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fertility treatments in the IVF unit of Belinson Hospital that require serial transvaginal ultrasound scans.
* Female age 18-43
* Normal pelvic anatomy
* Capable and willing to perform self vaginal ultrasound measurements.
* Ability to understand and sign the informed consent.
* Ability to read and understand instructions that are required for equipment use
* Ability to identify the uterus and ovaries on the device screen by the end of the training session.
* Patient can read and understand Hebrew or English

Exclusion Criteria:

* Known uterine malformations.
* Known ovarian pathologies.
* Known or suspected diminished ovarian reserve parameters (basal FSH> 10 IU/L, AFC <7 or serum AMH < 1ng/ml), unless 9 or more oocytes were aspirated in a previous ART cycle within the last 3 months.
* Presence of hydrosalpinx.
* Intraabdominal adhesions.
* Previous lower abdominal surgery.
* BMI >40
* Unable to use the trans-vaginal device.
* Subjects allergic to the ultrasound probe materials.
* Significant malposition of the ovaries.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incident of device related, or procedure related severe adverse events | 24 months
  The incidence of procedure related severe adverse events will be established, using reporting system for each individual subject enrolled in the study. The primary safety endpoint for each study subject is whether there is severe device- or procedure- related adverse events observed during the study. The resulting event rates will be established separately for the video guided and clinician guided modes of the device.
Comparison of device visualization of ovaries and uterus in a sagittal view to ground truth in each visit | 24 months
  The visualization of the ovaries and uterus in a sagittal view would be matched with the visualization of the ovaries and uterus derived by the ground truth (in-clinic ultrasound scan)

SECONDARY OUTCOMES:
Comparison of number of follicles >17 mm during the last IVF visit to ground truth | 24 months
  The number of ovarian follicles >17 mm at the last visit will be counted and matched with the number of ovarian follicles >17 mm at the last visit derived by the ground truth (in-clinic ultrasound scan)
Comparison of endometrium thickness during the last IVF visit to ground truth | 24 months
  The endometrium thickness at the last visit will be measured and matched with the endometrium thickness at the last visit derived by the ground truth (in-clinic ultrasound scan)

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van den Heuvel JF, Groenhof TK, Veerbeek JH, van Solinge WW, Lely AT, Franx A, Bekker MN. eHealth as the Next-Generation Perinatal Care: An Overview of the Literature. J Med Internet Res. 2018 Jun 5;20(6):e202. doi: 10.2196/jmir.9262. PMID 29871855
- [Result] Gerris J. Telemonitoring in IVF/ICSI. Curr Opin Obstet Gynecol. 2017 Jun;29(3):160-167. doi: 10.1097/GCO.0000000000000363. PMID 28362680
- [Result] Kalafat E, Mir I, Perry H, Thilaganathan B, Khalil A. Is home blood-pressure monitoring in hypertensive disorders of pregnancy consistent with clinic recordings? Ultrasound Obstet Gynecol. 2018 Oct;52(4):515-521. doi: 10.1002/uog.19094. Epub 2018 Sep 10. PMID 29786155
- [Result] Tucker KL, Bankhead C, Hodgkinson J, Roberts N, Stevens R, Heneghan C, Rey E, Lo C, Chandiramani M, Taylor RS, North RA, Khalil A, Marko K, Waugh J, Brown M, Crawford C, Taylor KS, Mackillop L, McManus RJ. How Do Home and Clinic Blood Pressure Readings Compare in Pregnancy? Hypertension. 2018 Sep;72(3):686-694. doi: 10.1161/HYPERTENSIONAHA.118.10917. PMID 30354754
- [Result] Moy FM, Ray A, Buckley BS, West HM. Techniques of monitoring blood glucose during pregnancy for women with pre-existing diabetes. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009613. doi: 10.1002/14651858.CD009613.pub3. PMID 28602020
- [Result] Raman P, Shepherd E, Dowswell T, Middleton P, Crowther CA. Different methods and settings for glucose monitoring for gestational diabetes during pregnancy. Cochrane Database Syst Rev. 2017 Oct 29;10(10):CD011069. doi: 10.1002/14651858.CD011069.pub2. PMID 29081069
- [Result] Romano M, Cesarelli M, D'Addio G, Mazzoleni MC, Bifulco P, Ferrara N, Rengo F. Telemedicine fetal phonocardiography surveillance: an italian satisfactory experience. Stud Health Technol Inform. 2010;155:176-81. PMID 20543326
- [Result] Kovacs F, Torok M, Horvath C, Balogh AT, Zsedrovits T, Nagy A, Hosszu G. A new, phonocardiography-based telemetric fetal home monitoring system. Telemed J E Health. 2010 Oct;16(8):878-82. doi: 10.1089/tmj.2010.0039. Epub 2010 Oct 6. PMID 20925563